CLINICAL TRIAL: NCT05340010
Title: Administration of Human Chorionic Gonadotrophin Before Secretory Transformation of Frozen-thawed Embryo Transfer Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCG in FET cycles
Record Dates: First submitted 2022-02-08; First posted 2022-04-21 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2021-12

CONDITIONS: hCG; FET; Frozen-thawed Embryo Transfe; Human Chorionic Gonadotrophin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCG group (Experimental): n Group 1 (hCG): participants will receive endometrial preparation with estrogen and an intramuscular hCG injection will before progesterone supplementation
  Interventions: Drug: Human Chorionic Gonadotrophin Intramuscular injection 10.000 IU
- control group (No Intervention): Group 2 (control): participants will receive the conventional endometrial preparation with estrogen followed by progesterone supplementation

INTERVENTIONS:
Drug: Human Chorionic Gonadotrophin Intramuscular injection 10.000 IU — From the 12th to 13th day of the cycle when endometrium reached the optimal thickness ≥8 mm, group 1 (hCG) will receive 10.000 IU hCG intramuscular injection in the morning then vaginal suppository progesterone 400 mg twice a day will be started in the afternoon
  Arms: HCG group

SUMMARY:
Successful embryo implantation is complicated process that requires synchrony between good-quality embryos and receptive endometrium. Human chorionic gonadotropin (hCG), is one of the initial embryonic signals and the major embryoendometrial relationship regulator. This study will be conducted to to investigate the role of parenteral hCG used for the transfer of cryopreserved- thawed embryos with HRT cycles in the outcome of artificially prepared frozen embryo transfer (FET) cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≤ 38 years.
* Normal 3D transvaginal ultrasound.
* At least two good quality embryos cryopreserved by vitrification.
* No GnRH agonists administration before FET cycle.

Exclusion Criteria

* Endometriosis.
* Uterine anomalies.
* Evidence of hydrosalpinx by hystrosalpingography or ultrasound.
* Evidence of immune disease, hematological or hormonal disorder.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 180 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Live birth delivery rate (LBR) | 7 months
  Number of live births beyond 28 weeks of gestational age to the total number of FET cycles

SECONDARY OUTCOMES:
Clinical pregnancy rate | 2 weeks after positive pregnancy test
  number of cases with observed gestational sac with embryonic heartbeat detected by ultrasound two weeks after positive pregnancy to the totoal number of frozen embryo transfer cycles.
Implantation rate | 2 weeks after positive pregnancy test
  proportion of the number of gestational sacs to the number of embryos transferred
Miscarriage rate | 20 weeks gestational age
  number of lost before the 20th week of gestation to the number of clinical pregnancies

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

REFERENCES:
- [Background] Licht P, Fluhr H, Neuwinger J, Wallwiener D, Wildt L. Is human chorionic gonadotropin directly involved in the regulation of human implantation? Mol Cell Endocrinol. 2007 Apr 15;269(1-2):85-92. doi: 10.1016/j.mce.2006.09.016. Epub 2007 Feb 14. PMID 17367920
- [Background] Tan H, Hu S; Qiongyu; Chen Y, Jin L, Wu C. The Effect of Intrauterine Administration of Human Chorionic Gonadotropin (hCG) Before Embryo Transfer During Assisted Reproductive Cycles: a Meta-Analysis of Randomized Controlled Trials. Geburtshilfe Frauenheilkd. 2019 Jul;79(7):713-722. doi: 10.1055/a-0837-3246. Epub 2019 Apr 1. PMID 31303659
- [Background] Gao M, Jiang X, Li B, Li L, Duan M, Zhang X, Tian J, Qi K. Intrauterine injection of human chorionic gonadotropin before embryo transfer can improve in vitro fertilization-embryo transfer outcomes: a meta-analysis of randomized controlled trials. Fertil Steril. 2019 Jul;112(1):89-97.e1. doi: 10.1016/j.fertnstert.2019.02.027. PMID 31277770
- [Background] Tesarik J, Hazout A, Mendoza C. Luteinizing hormone affects uterine receptivity independently of ovarian function. Reprod Biomed Online. 2003 Jul-Aug;7(1):59-64. doi: 10.1016/s1472-6483(10)61729-4. PMID 12930575
- [Background] Laokirkkiat P, Thanaboonyawat I, Boonsuk S, Petyim S, Prechapanich J, Choavaratana R. Increased implantation rate after intrauterine infusion of a small volume of human chorionic gonadotropin at the time of embryo transfer: a randomized, double-blind controlled study. Arch Gynecol Obstet. 2019 Jan;299(1):267-275. doi: 10.1007/s00404-018-4962-7. Epub 2018 Nov 17. PMID 30449012
- [Background] Shiotani M, Matsumoto Y, Okamoto E, Yamada S, Mizusawa Y, Furuhashi K, Ogata H, Ogata S, Kokeguchi S. Is human chorionic gonadotropin supplementation beneficial for frozen and thawed embryo transfer in estrogen/progesterone replacement cycles?: A randomized clinical trial. Reprod Med Biol. 2017 Apr 4;16(2):166-169. doi: 10.1002/rmb2.12023. eCollection 2017 Apr. PMID 29259465
- [Background] Deng L, Chen X, Blockeel C, Ye DS, Chen SL. Intramuscular injection of human chorionic gonadotropin prior to secretory transformation in patients undergoing frozen-thawed embryo transfer cycles. Reprod Biol Endocrinol. 2020 May 25;18(1):52. doi: 10.1186/s12958-020-00606-y. PMID 32450894
- [Result] Lawrenz B, Coughlan C, Melado L, Fatemi HM. The ART of frozen embryo transfer: back to nature! Gynecol Endocrinol. 2020 Jun;36(6):479-483. doi: 10.1080/09513590.2020.1740918. Epub 2020 Mar 18. PMID 32188299
- [Result] Ben-Meir A, Aboo-Dia M, Revel A, Eizenman E, Laufer N, Simon A. The benefit of human chorionic gonadotropin supplementation throughout the secretory phase of frozen-thawed embryo transfer cycles. Fertil Steril. 2010 Feb;93(2):351-4. doi: 10.1016/j.fertnstert.2009.02.027. Epub 2009 Apr 1. PMID 19342020
- [Result] Eftekhar M, Rahmani E, Eftekhar T. Effect of adding human chorionic gonadotropin to the endometrial preparation protocol in frozen embryo transfer cycles. Int J Fertil Steril. 2012 Oct;6(3):175-8. Epub 2012 Dec 17. PMID 24520435
- [Result] Jing S, Li XF, Zhang S, Gong F, Lu G, Lin G. Increased pregnancy complications following frozen-thawed embryo transfer during an artificial cycle. J Assist Reprod Genet. 2019 May;36(5):925-933. doi: 10.1007/s10815-019-01420-1. Epub 2019 Mar 29. PMID 30924053
- [Result] Hatoum I, Bellon L, Swierkowski N, Ouazana M, Bouba S, Fathallah K, Paillusson B, Bailly M, Boitrelle F, Alter L, Bergere M, Selva J, Wainer R. Disparities in reproductive outcomes according to the endometrial preparation protocol in frozen embryo transfer : The risk of early pregnancy loss in frozen embryo transfer cycles. J Assist Reprod Genet. 2018 Mar;35(3):425-429. doi: 10.1007/s10815-017-1078-0. Epub 2017 Nov 6. PMID 29110260
- [Result] Srivastava A, Sengupta J, Kriplani A, Roy KK, Ghosh D. Profiles of cytokines secreted by isolated human endometrial cells under the influence of chorionic gonadotropin during the window of embryo implantation. Reprod Biol Endocrinol. 2013 Dec 17;11:116. doi: 10.1186/1477-7827-11-116. PMID 24345207
- [Result] Makrigiannakis A, Vrekoussis T, Zoumakis E, Kalantaridou SN, Jeschke U. The Role of HCG in Implantation: A Mini-Review of Molecular and Clinical Evidence. Int J Mol Sci. 2017 Jun 19;18(6):1305. doi: 10.3390/ijms18061305. PMID 28629172
- [Result] Licht P, von Wolff M, Berkholz A, Wildt L. Evidence for cycle-dependent expression of full-length human chorionic gonadotropin/luteinizing hormone receptor mRNA in human endometrium and decidua. Fertil Steril. 2003 Mar;79 Suppl 1:718-23. doi: 10.1016/s0015-0282(02)04822-7. PMID 12620482